CLINICAL TRIAL: NCT03854370
Title: A Randomized Trial of Vaginal Prep Solutions to Reduce Bacteria Colony Counts in Patients Having a Vaginal Surgery
Brief Title: Vaginal Prep Solutions to Reduce Bacteria Colony Counts in Patients Having a Vaginal Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID impact on recruitment; challenges with enrollment
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 06612
Record Dates: First submitted 2019-01-18; First posted 2019-02-26 (Actual); Results first posted 2024-04-15 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Surgical Site Infection; Vaginal Surgery
Keywords: surgical prep; vaginal prep; baby shampoo
MeSH Terms: conditions — Surgical Wound Infection | interventions — Povidone-Iodine; chlorhexidine gluconate; Chlorhexidine

STUDY DESIGN:
Intervention Model Description: Randomized to 1 of 4 surgical prep agents
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and laboratory staff will not know which group cases have been assigned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Baby shampoo (Experimental): Baby shampoo used for surgical site prep
  Interventions: Other: Baby shampoo
- Peridex (Chlorhexidine) (Active Comparator): Peridex used for surgical site prep
  Interventions: Other: Peridex
- TechniCare (chloroxynel) (Active Comparator): TechniCare used for surgical site prep
  Interventions: Other: TechniCare
- Betadine (Povidone- iodine) (Active Comparator): Betadine used for surgical site prep
  Interventions: Other: Betadine

INTERVENTIONS:
Other: Baby shampoo — baby shampoo will be used to prepare the surgical site prior to incision
  Arms: Baby shampoo
Other: Betadine — Betadine (Povidone- iodine) will be used to prepare the surgical site prior to incision
  Other Names: Povidone- iodine
  Arms: Betadine (Povidone- iodine)
Other: Peridex — Peridex (Chlorhexidine) will be used to prepare the surgical site prior to incision
  Other Names: Chlorhexidine
  Arms: Peridex (Chlorhexidine)
Other: TechniCare — TechniCare (chloroxynel) will be used to prepare the surgical site prior to incision
  Other Names: chloroxynel
  Arms: TechniCare (chloroxynel)

SUMMARY:
This is a randomized trial comparing the effectiveness of 4 vaginal prep solutions (betadine, baby shampoo, TechniCare and Peridex) on reducing bacterial colony counts during surgery preparation. Women undergoing a vaginal surgery will be enrolled into the trial prior to surgery. Target sample size per group is 15 patients. During standard surgical prep, a vaginal swab will be taken to assess the initial colony counts for aerobic and anaerobic bacteria. After the initial swab, the incision point will be prepared using one of the prep 4 solutions (betadine, baby shampoo, TechniCare or Peridex). After a predefined 10 minutes, the area will be re-swabbed to determine pre-incision colony counts. A third swab will be collected after incision closure. Laboratory analyses for raw colony counts, sensitivities, identification (using MALDI-TOF) will be performed. The results are expected to show that there will be reduced colony counts at the pre-incision point with baby shampoo having the least reduction, followed by betadine and TechniCare, then Peridex. Patient reported outcomes for vaginal itching and burning as well as patient report of any treatment for vaginal infection will be collected by telephone at 2 days, 2 weeks and 1 month post-surgery.

DETAILED DESCRIPTION:
BACKGROUND AND LITERATURE REVIEW Antiseptic preparation for surgical incision sites has greatly reduced postoperative infections. However, surgical site infections (SSI) are still the leading cause of hospitalizations after surgery. With the application of antiseptic preparation, a reduction in bacterial counts follows. The rate at which the bacterial counts rise between preparation and incision may be of variation depending on the surgical antiseptic scrub.

Betadine (Povidone- iodine), Peridex (Chlorhexidine), baby shampoo and TechniCare (chloroxynel) are all surgical scrubs approved for the preparation of vaginal access surgeries. While there has been controversy on the use of Chlorohexidine for vaginal preparation surgery, due to its labeling as a cause for irritation, studies have shown that when 2-4% Chlorhexidine is used in the vaginal area there are little to no signs of irritation and the bacteria counts post incision are less than the bacterial counts for povidone iodine1,2. Baby shampoo can also be used as an effective antiseptic scrub with no irritation and no statistical difference in bacterial count reduction as compared to povidone-iodine3. Little research has been done to look at the antiseptic power of Chloroxynel in vaginal surgeries. However, when used as a root canal antiseptic it can reduce bacteria counts by 99.9%4. This is illustrative of its capability to reduce bacteria on a mucus membrane similar to the vagina.

There is literature that shows the antiseptic power of Betadine, Peridex, Baby shampoo and TechniCare for post-incisional bacteria counts, but little is known about the pre-incisional power of these scrubs for vaginal access surgeries.

SPECIFIC AIMS OR OBJECTIVES The aim of this study is to understand the power of vaginal surgical scrubs before incision. This will be done by collecting bacterial samples both before and 10 minutes after antiseptic preparation and after incision closure, along with follow-up data of irritation, infection post-surgery, and infection risk factors of each patient.

SIGNIFICANCE TO PATIENT, INSTITUTION, PROFESSION, OR ALL Vaginal preparation research provides benefitted knowledge to hospitals and physicians in the prevention of surgical site infections (SSI). This specific project will provide insight regarding the bacteria-eliminating power of four different surgical scrubs used on the vaginal mucous membrane, pre-incision. There is potential for this study to determine the most effective scrub for vaginal surgeries, as well as correlate pre-incisional bacterial counts and the post-procedure bacterial counts with likelihood of surgical site infections. The information collected from this study could benefit future patients and hospitals alike in terms of reducing the risk of SSI's. The risks of this study could be unidentified allergies to any of the surgical scrubs, or a loss of patient data. These are unlikely risks due to the protocol of the study.

METHODS This study will use block randomization. There will be four arms of the study one for each of the four surgical scrubs. There will be approximately 15 patients per arm. Patients undergoing vaginal surgeries will be recruited from Wright State Physicians Obstetrics and Gynecology. All procedures that require a vaginal incision will be included in the study, these being procedures like hysterectomies and reconstruction surgery. Non-incisional procedures like dilation and curettage will be excluded. Revision surgeries will also be excluded to decrease any complications. Patients who consent to the study will be given a ID and will be randomly assigned to one of the four arms. Patients will be excluded if an allergy to any of the scrubs is listed or found. Each recruited patient will be over the age of 18 with ability to provide consent.

Each patient will be given a standard prophylaxis 30 minutes before surgery. After prophylaxis administration and before surgical antiseptic preparation, a one minute swab will be taken of the vagina making sure to span the surface area of the vaginal canal with avoidance of the cervix. The swab will then be broken off into a tube labeled with the patient ID, date, and "pre-scrub". The patient will then undergo antiseptic preparation with the assigned surgical prep. A standard procedure of application will be done for each of the arms. Ten minutes after application, another swab will be taken using the same procedure as the "pre-scrub" swab. This swab will be broken off in a tube labeled with the patient ID, date, and "post-scrub"1. After incision closure, a third swab will be taken and will be labeled 'post-procedure'. The swabs will then be transported to CompuNet for analysis of aerobic, anaerobic bacteria and fungal colonies using Matrix Assisted Depolarization/Ionization Time of Flight mass spectrometry (MADI-TOF).

The data of colony counts will be collected from CompuNet. BMI, age, prophylaxis, postmenopausal information, diabetic information, smoking history, surgical duration, complication in surgery, and length of hospital stay will all be collected from patient records. No patient identifiers will be collected5. Patients will be followed up after surgery approximately two days, two weeks and a month after surgery to get information on irritation and/or surgical infection. This data will be collected either be phone call or at post-surgical follow-up appointment at Wright State Physicians. The South Hampton Grading Scheme for Surgical Wounds will be used to Quantify Each patients level of irritation and/or infection. The scale is a Zero to Five score, with Zero being no irritation or infection and Five being severe irritation or infection15.

One potential obstacle of this study could be recruitment of patients. Patients will not be given incentive for participation and will not acquire any direct benefit from the study. Another potential issue may arise from the size of the study; there may not be enough subjects recruited for each arm of the study to find a detectable and significant difference in the use of one surgical scrub over another.

Precautions will need to be taken for allergies. A recruited patient may not be aware of personal allergies to the surgical scrubs. This would put the patient at risk of harm if there was the potential for having an allergy to the assigned scrub. Since data will be collected from the patient's medical records, precautions will be taken to avoid loss of patient identifiers. All research investigators will only utilize the patients assigned research ID. This will both protect the patient and avoid bias.

ELIGIBILITY:
Inclusion Criteria:

* All procedures that require a vaginal incision will be included in the study, these being procedures like hysterectomies and reconstruction surgery.

Exclusion Criteria:

* Non-incisional procedures like dilation and curettage will be excluded.
* Revision surgeries will also be excluded to decrease any complications.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Towers, MD, Principal Investigator — Wright State Univeristy
Locations (1):
- Wright State Physicians, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on a case by case basis
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year after completion of the study
Access Criteria: Considered on a case by case basis

REFERENCES:
- [Background] Culligan PJ, Kubik K, Murphy M, Blackwell L, Snyder J. A randomized trial that compared povidone iodine and chlorhexidine as antiseptics for vaginal hysterectomy. Am J Obstet Gynecol. 2005 Feb;192(2):422-5. doi: 10.1016/j.ajog.2004.08.010. PMID 15695981
- [Background] Al-Niaimi A, Rice LW, Shitanshu U, Garvens B, Fitzgerald M, Zerbel S, Safdar N. Safety and tolerability of chlorhexidine gluconate (2%) as a vaginal operative preparation in patients undergoing gynecologic surgery. Am J Infect Control. 2016 Sep 1;44(9):996-8. doi: 10.1016/j.ajic.2016.02.036. Epub 2016 May 24. PMID 27234011
- [Background] Garcia GA, Nguyen CV, Yonkers MA, Tao JP. Baby Shampoo Versus Povidone-Iodine or Isopropyl Alcohol in Reducing Eyelid Skin Bacterial Load. Ophthalmic Plast Reconstr Surg. 2018 Jan/Feb;34(1):43-48. doi: 10.1097/IOP.0000000000000850. PMID 28072611
- [Background] Lewis LA, Lathi RB, Crochet P, Nezhat C. Preoperative vaginal preparation with baby shampoo compared with povidone-iodine before gynecologic procedures. J Minim Invasive Gynecol. 2007 Nov-Dec;14(6):736-9. doi: 10.1016/j.jmig.2007.05.010. PMID 17980335
- [Background] Schafer E, Bossmann K. Antimicrobial efficacy of chloroxylenol and chlorhexidine in the treatment of infected root canals. Am J Dent. 2001 Aug;14(4):233-7. PMID 11699743
- [Background] American College of Obstetricians and Gynecologists Women's Health Care Physicians; Committee on Gynecologic Practice. Committee Opinion No. 571: Solutions for surgical preparation of the vagina. Obstet Gynecol. 2013 Sep;122(3):718-20. doi: 10.1097/01.AOG.0000433982.36184.95. PMID 23963423
- [Background] Van Wicklin SA. Preoperative vaginal preps with chlorhexidine gluconate solution. Am J Obstet Gynecol. 2006 Aug;195(2):624; author reply 625. doi: 10.1016/j.ajog.2005.11.002. Epub 2006 Apr 21. No abstract available. PMID 16890564
- [Background] Vorherr H, Ulrich JA, Messer RH, Hurwitz EB. Antimicrobial effect of chlorhexidine on bacteria of groin, perineum and vagina. J Reprod Med. 1980 Apr;24(4):153-7. PMID 7373599
- [Background] Aly R, Maibach HI. Comparative antibacterial efficacy of a 2-minute surgical scrub with chlorhexidine gluconate, povidone-iodine, and chloroxylenol sponge-brushes. Am J Infect Control. 1988 Aug;16(4):173-7. doi: 10.1016/0196-6553(88)90029-6. PMID 3189943
- [Background] Culver DH, Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG, Banerjee SN, Edwards JR, Tolson JS, Henderson TS, et al. Surgical wound infection rates by wound class, operative procedure, and patient risk index. National Nosocomial Infections Surveillance System. Am J Med. 1991 Sep 16;91(3B):152S-157S. doi: 10.1016/0002-9343(91)90361-z. PMID 1656747
- [Background] Faro C, Faro S. Postoperative pelvic infections. Infect Dis Clin North Am. 2008 Dec;22(4):653-663. doi: 10.1016/j.idc.2008.05.005. PMID 18954757
- [Background] Kjolhede P, Halili S, Lofgren M. Vaginal cleansing and postoperative infectious morbidity in vaginal hysterectomy. A register study from the Swedish National Register for Gynecological Surgery. Acta Obstet Gynecol Scand. 2011 Jan;90(1):63-71. doi: 10.1111/j.1600-0412.2010.01023.x. Epub 2010 Nov 26. PMID 21275917
- [Background] Steiner HL, Strand EA. Surgical-site infection in gynecologic surgery: pathophysiology and prevention. Am J Obstet Gynecol. 2017 Aug;217(2):121-128. doi: 10.1016/j.ajog.2017.02.014. Epub 2017 Feb 14. PMID 28209490
- [Background] Bailey IS, Karran SE, Toyn K, Brough P, Ranaboldo C, Karran SJ. Community surveillance of complications after hernia surgery. BMJ. 1992 Feb 22;304(6825):469-71. doi: 10.1136/bmj.304.6825.469. PMID 1547415

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Baby Shampoo | Peridex (Chlorhexidine) | TechniCare (Chloroxynel) | Betadine (Povidone- Iodine)
Started | 9 | 9 | 7 | 10
Completed | 8 | 8 | 6 | 9
Not Completed | 1 | 1 | 1 | 1
Not completed — samples not collected | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baby Shampoo | Peridex (Chlorhexidine) | TechniCare (Chloroxynel) | Betadine (Povidone- Iodine) | Total
Number analyzed (Participants) | 8 | 8 | 6 | 9 | 31
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 39.4 (8.7) | 44.9 (8.7) | 44.0 (10.2) | 46.8 (17.3) | 43.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 6 | 9 | 31
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 6 | 9 | 31
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.7 (1.5) | 31.0 (7.3) | 27.0 (2.6) | 28.0 (7.1) | 30.5 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Vaginal Colony Counts (Anaerobic)
Description: anaerobic culture colony counts - change in anaerobic colony counts from prior to surgical prep to 10 minutes after surgical prep
Time Frame: 2 timepoints: prior to surgical prep, and 10 min after surgical prep
Measure: Count of Participants; unit: Participants
Arm/Group | Baby Shampoo | Peridex (Chlorhexidine) | TechniCare (Chloroxynel) | Betadine (Povidone- Iodine)
Number analyzed (Participants) | 8 | 8 | 6 | 9
Participants
  Prior to surgical scrub: # participants with positive cultures | 6 | 8 | 6 | 8
  Prior to surgical scrub: # participants with negative cultures | 2 | 0 | 0 | 1
  Post surgical scrub: # participants with positive cultures | 4 | 5 | 1 | 3
  Post surgical scrub: # participants with negative cultures | 4 | 3 | 5 | 6
Statistical Analysis 1: Comparison: Baby Shampoo vs Peridex (Chlorhexidine) vs TechniCare (Chloroxynel) vs Betadine (Povidone- Iodine); Comparison of all four groups prior to surgical scrub; Test type: Superiority; p = 0.23, Chi-squared
Statistical Analysis 2: Comparison: Baby Shampoo vs Betadine (Povidone- Iodine); Comparison of baby shampoo versus iodine post surgical scrub; Test type: Superiority; p = 0.31, Fisher Exact
Statistical Analysis 3: Comparison: Peridex (Chlorhexidine) vs Betadine (Povidone- Iodine); Comparison of Chlorhexidine versus iodine post surgical scrub; Test type: Superiority; p = .35, Fisher Exact
Statistical Analysis 4: Comparison: TechniCare (Chloroxynel) vs Betadine (Povidone- Iodine); Comparison of chloroxynel versus iodine post surgical scrub; Test type: Superiority; p = .61, Fisher Exact

2. Primary Outcome: Vaginal Colony Counts (Aerobic)
Description: aerobic culture colony counts - change in aerobic colony counts from prior to surgical prep to 10 minutes after surgical prep
Time Frame: 2 timepoints: prior to surgical prep, and 10 min after surgical prep
Measure: Count of Participants; unit: Participants
Arm/Group | Baby Shampoo | Peridex (Chlorhexidine) | TechniCare (Chloroxynel) | Betadine (Povidone- Iodine)
Number analyzed (Participants) | 8 | 8 | 6 | 9
Participants
  Prior to surgical scrub: # participants with positive cultures | 6 | 8 | 5 | 9
  Prior to surgical scrub: # participants with negative cultures | 2 | 0 | 1 | 0
  Post surgical scrub: # participants with positive cultures | 5 | 4 | 0 | 1
  Post surgical scrub: # participants with negative cultures | 3 | 4 | 6 | 8
Statistical Analysis 1: Comparison: Baby Shampoo vs Peridex (Chlorhexidine) vs TechniCare (Chloroxynel) vs Betadine (Povidone- Iodine); comparison of all four groups prior to surgical scrub; Test type: Superiority; p = .59, Chi-squared
Statistical Analysis 2: Comparison: Baby Shampoo vs Betadine (Povidone- Iodine); Comparison of baby shampoo versus iodine post surgical scrub; Test type: Superiority; p = .05, Fisher Exact
Statistical Analysis 3: Comparison: Peridex (Chlorhexidine) vs Betadine (Povidone- Iodine); Comparison of chlorhexidine versus iodine post surgical scrub; Test type: Superiority; p = .13, Fisher Exact
Statistical Analysis 4: Comparison: TechniCare (Chloroxynel) vs Betadine (Povidone- Iodine); Comparison of chloroxynel versus iodine at post surgical scrub; Test type: Superiority; p = 0.99, Fisher Exact

3. Secondary Outcome: Vaginal Colony Counts (Fungal)
Description: fungal culture colony counts - change in fungal colony counts from prior to surgical prep to 10 minutes after surgical prep
Time Frame: 2 timepoints: prior to surgical prep, and 10 min after surgical prep
Measure: Count of Participants; unit: Participants
Arm/Group | Baby Shampoo | Peridex (Chlorhexidine) | TechniCare (Chloroxynel) | Betadine (Povidone- Iodine)
Number analyzed (Participants) | 8 | 8 | 6 | 9
Participants
  Prior to surgical scrub: # participants with positive culture | 1 | 0 | 1 | 0
  Prior to surgical scrub: # participants with negative culture | 7 | 8 | 5 | 9
  Post surgical scrub: # participants with positive culture | 0 | 0 | 0 | 0
  Post surgical scrub: # participants with negative culture | 8 | 8 | 6 | 9
Statistical Analysis 1: Comparison: Baby Shampoo vs Peridex (Chlorhexidine) vs TechniCare (Chloroxynel) vs Betadine (Povidone- Iodine); Comparison of all four groups prior to surgical scrub; Test type: Superiority; p = 0.45, Chi-squared
Statistical Analysis 2: Comparison: Baby Shampoo vs Betadine (Povidone- Iodine); Comparison of baby shampoo versus iodine post surgical scrub; Test type: Superiority; p = 0.99, Fisher Exact — all groups were negative for cultures
Statistical Analysis 3: Comparison: Peridex (Chlorhexidine) vs Betadine (Povidone- Iodine); Comparison of chlorhexidine versus iodine at post surgical scrub; Test type: Superiority; p = 0.99, Fisher Exact — All groups had negative cultures
Statistical Analysis 4: Comparison: TechniCare (Chloroxynel) vs Betadine (Povidone- Iodine); Comparison of chloroxynel versus iodine at post surgical scrub; Test type: Superiority; p = 0.99, Fisher Exact — All groups had negative cultures

4. Secondary Outcome: Vaginal Colony Counts (Anaerobic)
Description: Change in anaerobic culture colony counts from 10 min after surgical prep (prior to incision) to post-procedure (incision closure)
Time Frame: 2 timepoints: 10 min after surgical prep (prior to incision), and after incision closure
Measure: Count of Participants; unit: Participants
Arm/Group | Baby Shampoo | Peridex (Chlorhexidine) | TechniCare (Chloroxynel) | Betadine (Povidone- Iodine)
Number analyzed (Participants) | 8 | 8 | 6 | 9
Participants
  Post surgical prep: # participants with positive cultures | 4 | 5 | 1 | 3
  Post surgical prep: # participants with negative cultures | 4 | 3 | 5 | 6
  Post procedure: # participants with positive cultures | 3 | 3 | 3 | 4
  Post procedure: # participants with negative cultures | 5 | 5 | 3 | 5
Statistical Analysis 1: Comparison: Baby Shampoo vs Betadine (Povidone- Iodine); Comparison of baby shampoo versus iodine at post procedure; Test type: Superiority; p = 0.61, Fisher Exact
Statistical Analysis 2: Comparison: Peridex (Chlorhexidine) vs Betadine (Povidone- Iodine); Comparison of chlorhexidine versus iodine at post procedure; Test type: Superiority; p = 0.99, Fisher Exact
Statistical Analysis 3: Comparison: TechniCare (Chloroxynel) vs Betadine (Povidone- Iodine); Comparison of chloroxynel versus iodine at post procedure; Test type: Superiority; p = 0.99, Fisher Exact

5. Secondary Outcome: Vaginal Colony Counts (Aerobic)
Description: Change in aerobic culture colony counts from 10 min after surgical prep (prior to incision) to post-procedure (incision closure)
Time Frame: 2 timepoints: 10 min after surgical prep (prior to incision), and after incision closure
Measure: Count of Participants; unit: Participants
Arm/Group | Baby Shampoo | Peridex (Chlorhexidine) | TechniCare (Chloroxynel) | Betadine (Povidone- Iodine)
Number analyzed (Participants) | 8 | 8 | 6 | 9
Participants
  Post surgical scrub: # participants with positive cultures | 5 | 4 | 0 | 1
  Post surgical scrub: # participants with negative cultures | 3 | 4 | 6 | 8
  Post procedure: # participants with positive cultures | 4 | 1 | 0 | 2
  Post procedure: # participants with negative cultures | 4 | 7 | 6 | 7
Statistical Analysis 1: Comparison: Baby Shampoo vs Betadine (Povidone- Iodine); Comparison of baby shampoo versus iodine at post procedure; Test type: Superiority; p = 0.32, Fisher Exact
Statistical Analysis 2: Comparison: Peridex (Chlorhexidine) vs Betadine (Povidone- Iodine); Comparison of chlorhexidine versus iodine at post procedure; Test type: Superiority; p = 0.99, Fisher Exact
Statistical Analysis 3: Comparison: TechniCare (Chloroxynel) vs Betadine (Povidone- Iodine); Comparison of chloroxynel versus iodine at post procedure; Test type: Superiority; p = 0.50, Fisher Exact

6. Secondary Outcome: Vaginal Colony Counts (Fungal)
Description: Change in fungal culture colony counts from 10 min after surgical prep (prior to incision) to post-procedure (incision closure)
Time Frame: 2 timepoints: 10 min after surgical prep (prior to incision), and after incision closure
Measure: Count of Participants; unit: Participants
Arm/Group | Baby Shampoo | Peridex (Chlorhexidine) | TechniCare (Chloroxynel) | Betadine (Povidone- Iodine)
Number analyzed (Participants) | 8 | 8 | 6 | 9
Participants
  Post surgical scrub: # participants with positive cultures | 0 | 0 | 0 | 0
  Post surgical scrub: # participants with negative cultures | 8 | 8 | 6 | 9
  Post procedure: # participants with positive cultures | 0 | 0 | 0 | 0
  Post procedure: # participants with negative cultures | 8 | 8 | 6 | 9
Statistical Analysis 1: Comparison: Baby Shampoo vs Betadine (Povidone- Iodine); Comparison of baby shampoo versus iodine at post procedure; Test type: Superiority; p = 0.99, Fisher Exact — All groups had negative cultures
Statistical Analysis 2: Comparison: Peridex (Chlorhexidine) vs Betadine (Povidone- Iodine); comparison of chlorhexidine versus iodine at post procedure; Test type: Superiority; p = 0.99, Fisher Exact — All groups had negative cultures
Statistical Analysis 3: Comparison: TechniCare (Chloroxynel) vs Betadine (Povidone- Iodine); Comparison of chloroxynel versus iodine at post procedure; Test type: Superiority; p = 0.99, Fisher Exact — All groups had negative cultures

ADVERSE EVENTS:
Time Frame: 1 month post operation
Arm/Group | Baby Shampoo | Peridex (Chlorhexidine) | TechniCare (Chloroxynel) | Betadine (Povidone- Iodine)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/6 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/6 | 0/9

LIMITATIONS AND CAVEATS:
This study does have significant limitations which make application to all vaginal surgeries difficult. The small sample size increases the risk of bias so these results should be interpreted with caution. We experienced several challenges that impacted our enrollment of patients into the study including the cancellation of elective surgeries during the COVID-19 pandemic, and several periods when PCMX was not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT03854370/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT03854370/ICF_001.pdf